CLINICAL TRIAL: NCT05889273
Title: An Open-label Extension Study to Investigate Safety and Tolerability of ML-004 in Adolescents and Adults With Autism Spectrum Disorders (ASD).
Brief Title: ML-004 Open-Label Extension Study in Adults and Adolescents With Autism Spectrum Disorders (ASD)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: MapLight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML-004-003
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism; Autism Spectrum Disorder; Social Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ML-004 (IR)/(ER) tablet (Experimental): ML-004 is a bilayer immediate-release (IR)/extended-release (ER, gastroretentive) oral tablet formulation. ML-004 is taken orally once daily and provided as a tablet in two dose strengths of 12 mg (3 mg IR/9 mg ER) and 24 mg tablet (6 mg IR/18 mg ER). Dose levels for this study are 12 mg (provided as one 12 mg tablet), 24 mg (one 24 mg tablet), 48 mg (two 24 mg tablets), and 72 mg (three 24 mg tablets).
  Interventions: Drug: ML-004 (IR)/(ER) tablet

INTERVENTIONS:
Drug: ML-004 (IR)/(ER) tablet — Participants will receive ML-004 once daily.

SUMMARY:
ML-004-003 is a multi-center, open-label extension study that will enroll approximately 120 adolescent and adult subjects with ASD that have completed study ML-004-002. The primary objective of the study will be to evaluate the safety of ML-004 in subjects with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Has completed Study ML-004-002 within the past 90 days
* Age 12 years to 46 years at screening
* Has a designated care/study partner who can reliably report on symptoms
* Has a diagnosis of Autism Spectrum Disorder (ASD)
* Has a body mass index (BMI) ≥18 kg/m²
* Psychoactive medications and adjunctive therapies stable for 4 weeks prior to screening
* Must be able to swallow study medication

Exclusion Criteria:

* Has Rett syndrome or Child Disintegrative Disorder
* History of epilepsy without current adequate control, or any seizure in the 6 months preceding screening
* Has a positive response to C-SSRS questions 4 and/or 5, or is a significant risk for suicidal behavior
* Has a clinical history of uncontrolled or severe hypertension
* If female, is pregnant or lactating

Ages: 12 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of treatment-emergent adverse events (TEAEs). | Baseline up to Day 362

SECONDARY OUTCOMES:
Frequency of occurrence of Serious Adverse Events (SAEs) | Baseline up to Day 362
Frequency of occurrence of TEAEs leading to discontinuation. | Baseline up to Day 362
Frequency of occurrence of TEAEs arising from clinically important changes in other safety assessments. | Baseline up to Day 362
Frequency of occurrence of suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale. | Baseline up to Day 362

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Cortica Healthcare, Glendale, California
  - NRC Research Institute, Orange, California
  - Yale Child Study Center, New Haven, Connecticut
  - The Children's Research Institute, Washington D.C., District of Columbia
  - Abba Medical Group, Miami, Florida
  - APG Research, LLC, Orlando, Florida
  - University of South Florida Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - University of Missouri, Thompson Center for Autism & Neurodevelopment, Columbia, Missouri
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Suburban Research Associates, Media, Pennsylvania
  - BioBehavioral Research of Austin, Austin, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
- Australia (2):
  - Brain and Mind Centre, Camperdown, New South Wales
  - The Royal Children's Hospital, Murdoch Children's Research Institute, Parkville, Victoria
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ML-004-002 — https://clinicaltrials.gov/ct2/show/NCT05081245?term=ML-004&draw=2&rank=1